CLINICAL TRIAL: NCT06286449
Title: Identification of Cellular and Molecular Mechanisms Involved in the Pathophysiology of Alcohol Use Disorder by Examination of Cerebrospinal Fluid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSV_AUD
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Spinal Puncture

STUDY DESIGN:
Intervention Model Description: The intervention in this study consists of a spinal tap that all study participants undergo. We are comparing biomarkers in cerebrospinal fluid collected from either participants with Alcohol Use Disorder or from healthy controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alcohol Use Disorder cohort and Healthy controls cohort (Other): Alcohol Use Disorder Cohort The intervention, which all participants from both cohorts undergo, consists of a spinal tap, in which 35 ml of cerebrospinal fluid is collected for further analysis and comparison between a cohort consisting of healthy controls. Study participants with Alcohol Use Disorder (AUD) are recruited from other previous or ongoing clinical trials performed within the research group: NordAlc (PI Andrea de Bejczy), IV-ASA (PI Bo Söderpalm), GlycinA (PI Bo Söderpalm) and COMB (PI Bo Söderpalm).
  Healthy controls cohort The intervention, which all participants from both cohorts undergo, consists of a spinal tap, in which 35 ml of cerebrospinal fluid is collected for further analysis and comparison between a cohort consisting of participants with Alcohol Use Disorder. Healthy controls will be continuously recruited via advertisements in media, and onsite at the Sahlgrenska University Hospital and the University of Gothenburg
  Interventions: Other: Spinal tap

INTERVENTIONS:
Other: Spinal tap — A spinal tap is performed on all enrolled study participants that meet the eligibility criteria
  Other Names: Lumbar puncture

SUMMARY:
BACKGROUND

The brain and spinal cord are enveloped by cerebrospinal fluid (CSF), which extends down to the base of the spine, a few centimeters below the termination of the spinal cord. Here, it can be collected through a minor needle puncture. This procedure enables the gathering of information about otherwise concealed molecular and cellular processes in the brain. Analyzing various specific molecules in the CSF has yielded crucial insights into the underlying mechanisms of many neurological and psychiatric disorders, such as multiple sclerosis (MS) and dementia, significantly enhancing the prospects for its treatment. However, for several brain disorders, including Alcohol Use Disorder (AUD) and substance use disorders, CSF studies are absent. AUD, a brain disease affecting the reward system, is characterized by an inability to limit alcohol consumption. High levels of alcohol intake, as seen in AUD, are a leading cause of morbidity and premature mortality. Yet, there is a lack of effective medications for its treatment. Analyzing molecules in CSF, believed to be significant for the development and maintenance of AUD, could enhance the development of effective pharmacological treatments. At present, there are no CSF studies on individuals with AUD, that explore the underlying mechanisms of the disease. Additionally, several CSF studies lack a representative control group of truly healthy controls (i.e. have not presented any neurological or psychiatric symptoms), which is crucial for drawing accurate conclusions.

OBJECTIVE

Sub-study 1 aims to collect CSF from individuals with AUD across various ages to analyze brain molecules that contribute to the development and maintenance of the disease.

Sub-study 2 aims to gather CSF from healthy controls across various ages to study molecules involved in neurological and psychiatric conditions, including AUD, substance dependency, brain inflammation, and narcolepsy. The goal is to create a reference group of CSF from healthy controls for comparison with CSF collected from individuals with the aforementioned conditions.

We hypothesize that levels of certain molecules, such as dopamine, differ between healthy controls and those with e.g. AUD. This study may provide insights into cellular and molecular mechanisms underlying brain disorders, which is in turn crucial for developing new, effective treatments.

Sub-study 3 will examine how the incubation of nerve cells in CSF collected in sub-study 1 and 2 affects their excitability and ability to form new synapses, essential for communication in the brain.

We hypothesize that the excitability and synaptogenesis of nerve cells will vary depending on whether they are incubated in CSF from neurologically and psychiatrically healthy individuals versus those with AUD, substance use disorders, brain inflammation, and narcolepsy. Understanding how CSF composition influences brain function in these conditions could be instrumental in creating new therapeutic drugs.

METHODS

Individuals with AUD, as well as psychiatrically and neurologically healthy volunteers, will be successively recruited for CSF collection and analyses. Recruitment will be performed through media advertisements and posters within healthcare facilities (The Sahlgrenska University Hospital) and the University of Gothenburg. Additional participants will be recruited from parallel research projects performed within the group (IV-ASA BO10 dnr: 2019-04120, COMB BO8 dnr 431-18, GlycinA BO5 dnr 806-14, PI Bo Söderpalm and NordAlc BO9 dnr: 430-18, PI Andrea de Bejczy) CSF will be obtained through lumbar puncture (spinal tap), a procedure where a thin needle is inserted below the end of the spinal cord. Local anesthesia will be administered in order to mitigate potential discomfort. The lumbar puncture will be performed by an experienced physician, minimizing the risk of injury. Blood samples will also be collected to correlate molecule levels in CSF with those in the blood. Participants will be interviewed about their medical history including their alcohol consumption, and a comprehensive medical examination will be performed.

SIGNIFICANCE

CSF studies offers unique insights into the cellular and molecular processes within the brain. This approach has been utilized for exploring the mechanisms behind several psychiatric and neurological disorders, but not for certain brain diseases like AUD. AUD inflicts significant suffering for affected individuals, contributes to high mortality rates, and imposes considerable burdens on the society. Moreover, a deeper understanding of the cellular and molecular underpinnings of brain diseases such as AUD, can facilitate the development of novel, more effective medications for its treatment.

ELIGIBILITY:
Inclusion Criteria:

The study participant:

1. has given his/her written and oral informed consent to participate in the study
2. presents a breath alcohol concentration (BrAC) below 10mg% (10mg/dl) at the study visit

Exclusion Criteria:

The study participant:

1. is pregnant or breastfeeding
2. has an ongoing neurological or psychiatric disease except for Alcohol Use Disorder
3. has an ongoing or previous disease that affects either the safety of the study participant following a spinal tap or the outcome measures of the study
4. currently uses (within 30 days of enrollment) medication that affects either the safety of the study participant following a spinal tap or the outcome measures of the study
5. currently uses (within 30 days of enrollment) medications for the treatment of Alcohol Use Disorder or alcohol abstinence that affects the mesolimbic dopamine system
6. currently uses (within 30 days of enrollment) dietary supplements, including energy drinks, that may affect the safety for the study participant following a spinal tap or may have an impact on the outcome measures

8. currently and frequently uses (within 1 year of enrollment) drugs of abuse other than alcohol and nicotine.

9. participates in another interventional clinical trial within 30 days of enrollment

10. has a local infection or a tattoo in the lower back region

11. anatomical anomalies in the lower spine region, e.g. following prior spine surgery, that obstructs the procedure of a spinal tap

12. has prior history of allergic reactions to local anaesthetics

13. presents pathological findings during medical examination that may affect the safety for the study participant following a spinal tap or the outcome measures

14. is considered to be unfit for study participation for other reasons than stated above

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CSF-DA levels | 3 years
  Levels of dopamine in the cerebrospinal fluid

IPD SHARING:
Plan to Share IPD: No
The ethical approval does not allow us to share individual patient data, but only data presented on a group level, so that no individual patient can be identified.